CLINICAL TRIAL: NCT04615065
Title: Acutelines: a Large Biobank Aiming to Improve Early Recognition of Acute Diseases, Contribute to the Development of Personalized Medicine and Optimize Short- and Long-term Outcome
Brief Title: Acutelines: a Large Data-/Biobank of Acute and Emergency Medicine
Acronym: Acutelines
Status: Recruiting | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: 201900635
Record Dates: First submitted 2020-10-18; First posted 2020-11-04 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Acute Disease; Sepsis; Pneumonia; Frailty; Complication of Treatment; Pulmonary Embolism; Thrombosis; Acute Kidney Injury; Electrolyte Disturbance; Hemorrhage; Shock; Polypharmacy; Intoxication by Drug; Emergencies; Urinary Tract Infections; Skin Infection; Syncope; Anaphylaxis; Dyspnea
Keywords: Acute disease; Sepsis; Emergency Medical Service (EMS); Outcome; Precision medicine; Personalized medicine; Emergency medicine; Multidisciplinary; General practitionar; Pharmacy; Hospitalization; Health insurance; Mortality; Quality of life (QoL); Overcrowding; Patient logistics; Point-of-care ultrasound (POCUS); Helicopter Emergency Medical Service (HEMS); Biobank; Databank; Electrophysiological waveforms; Electrocardiogram (ECG); Plethysmogram
MeSH Terms: conditions — Acute Disease; Sepsis; Pneumonia; Frailty; Pulmonary Embolism; Thrombosis; Acute Kidney Injury; Hemorrhage; Shock; Emergencies; Urinary Tract Infections; Cellulitis; Syncope; Anaphylaxis; Dyspnea; Crowding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Biomaterials will be collected from:
  * Patients triaged as one of highest two triage categories (red or orange) according to the Manchester triage system;
  * Patients with shock;
  * Patients with a suspicion of sepsis (based on physicians' judgement, Sepsis-2 or Sepsis-3 criteria).
  Biomaterials to be collected are serum, plasma (EDTA), plasma (Lithium heparin), PAXGene RNA, buffy coat (from EDTA), urine, feces, hair
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Research in acute care faces many challenges, including enrollment challenges, legal limitations in data sharing, limited funding, and lack of singular ownership of the domain of acute care. To overcome some of these challenges, the Center of Acute Care of the University Medical Center Groningen in the Netherlands, has established a de novo data-, image- and biobank named "Acutelines". Acutelines is initiated to improve recognition and treatment of acute diseases and obtain insight in the consequences of acute diseases, including factors predicting its outcome. Thereby, Acutelines contributes to development of personalized treatment and improves prediction of patient outcomes after an acute admission.

DETAILED DESCRIPTION:
Acutelines is a prospective biobank including patients with a broad spectrum of acute conditions. Its aim is to facilitate interdisciplinary research on the etiology and development of acute diseases with the aid of systematically collected biomaterials and medical data over various timepoints, both during the course of the patient's disease and after recovery. Clinical data, imaging data and biomaterial (i.e. blood, urine, feces, hair) are collected for patients presenting to the Emergency Department (ED) with a broad range of acute disease presentations. A deferred consent procedure (by proxy), is in place to allow collecting data and biomaterials prior to obtaining written consent. The digital infrastructure in place and the software used ensures automated capturing of all bed-side monitoring data (i.e. electrophysiological waveforms, vital parameters), and the secure importation of data from other sources, such as the electronic health records of the hospital, ambulance and general practitioner, municipal registration, health insurance companies and pharmacy. Follow up data are collected for all included patients during the first 72-hours of their hospitalization and 3-months, 1-year, 2-years and 5 years after their ED visit.

Data and materials to be collected includes:

* Demographic and health data (i.e. [experiences] health, quality of life, functional status)
* Medical history (i.e. co-morbidity, intoxications, medication use)
* Admission reason to emergency department
* Physical examination and vital parameters
* Clinical diagnostic data (i.e. [point-of-care] ultrasound, X-ray, CT-scan, laboratory results)
* Electrophysiological waveforms (i.e. electrocardiogram [ECG], plethysmography)
* Biomaterials
* Treatment (i.e. medication use, non-pharmacological treatment, treatment decisions, length-of-stay in hospital, admission to intensive care unit [ICU])

ELIGIBILITY:
Inclusion Criteria, at least one of the following:

* Triaged as one of highest two triage categories (red or orange) according to the Manchester triage system;
* Triaged as the third highest triage category (yellow) and arrival by EMS of Helicopter Emergency Medical Service (HEMS;
* Shock
* Suspicion of sepsis (based on either physicians' suspicion, Sepsis-2 or Sepsis-3 criteria)
* Acute kidney injury (AKI)
* Anaphylactic reaction
* Syncope
* Intoxication
* Thrombosis
* Pulmonary embolism
* Bleeding while using anti-coagulant drugs
* Gastro-intestinal bleeding
* Electrolyte disturbance

Exclusion Criteria:

* Referred for organ transplantation as recipient
* Transfer from other hospital
* Accidental contact patient material (i.e. internal work-related accident)

While data- and imaging will be collected from all these patients, biomaterials will only be collected from patients fulfilling the first criterion (i.e. triaged as one of highest two triage categories [red or orange] according to the Manchester triage system) and from patients with shock or a suspicion of sepsis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to the emergency room for emergency medicine, internal medicine [including sub-specializations as allergology, acute medicine, oncology, hematology, infectiology, nephrology, vascular medicine, geriatric medicine], pulmonology, gastro-enterology and rheumatology.
Sampling Method: Non-Probability Sample
Enrollment: 35000 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2030-09-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
Mortality (time and cause) | Until the death of death from any cause, up to 50 years
  Mortality will be retrieved from the electronic health records (EHR) from the hospital and municipal registration. The cause of death will be retrieved from the EHR from the hospital, general practitioner and Dutch statistics' office (CBS).
Katz ADL-6 (functioning) | Up to 1 year
  Katz ADL-6 (0-6, fully dependent-independent)
World Health Organization (WHO) performance status (functioning) | Up to 1 year
  World Health Organization (WHO) performance status (0-4, normal performance-bedridden)
Karnofsky performance score (functioning) | Up to 1 year
  Karnofsky performance score (10-100, moribund-normal performance)
Utrecht Activity List (daily activities) | Up to 1 year
  Utrecht Activity List (UAL; hours/week spend on (a) paid work, (b) education, (c) household, (d) running errands, (e) unpaid work, (f) sport, (g) hobbies, (h) other use of leisure time )
Short QUestionnaire to ASsess Health-enhancing physical activity (daily activities) | Up to 1 year
  Short QUestionnaire to ASsess Health-enhancing physical activity (SQUASH; minutes/week and intensity of activity spend (a) commuting, (b) at work, (c) household activities and (d) leisure time; increased score corresponds with increased physical activity)
Quality of Life and experienced symptoms | Up to 1 year
  EuroQol-5D (EQ5D; simple descriptive profile and a single index value for health status; higher values corresponding with better health) with visual analogue scale (VAS; 0-100, worse-best experienced health)
Experienced somatic symptoms | Up to 1 year
  Patient Health Questionnaire-15 (PHQ-15; 0-30, minimal-high somatic symptom severity)
Fatigue | Up to 1 year
  Piper Fatigue Scale-12 (PFS-12; 0-10, higher scores reflect more fatigue among four subscales (a) behavior, (b) affect, (c) sensory, (d) cognition)
Patient Health Questionnaire-2 (mental health) | Up to 1 year
  Patient Health Questionnaire-2 (PHQ-2; 0-6, higher score corresponds to reduced mental health)
Patient Health Questionnaire-9 (mental health) | Up to 1 year
  Patient Health Questionnaire-9 (PHQ-9; 0-4 no depressive symptoms, 5-9 mild depressive symptoms, 10-14 moderate depressive symptoms, 15-19 moderately severe depressive symptoms, 20-27 severe depressive symptoms)
Geriatric Depression scale-15 (mental health) | Up to 1 year
  Geriatric Depression scale-15 (GDS-15; 0-4 no depressive symptoms, 5-10 mild depressive symptoms, 11-15 depressive symptoms)
Patient satisfaction | Up to 1 year
  Patient Satisfaction Questionnaire Short-form (PSQ-18; measuring general satisfaction, technical quality, interpersonal manner, communication, financial aspects, time spent with doctor, and accessibility and convenience; scored per domain, with lower scores corresponding with higher satisfaction)
Decision making | Up to 1 year
  Outcome prioritization tool (OPT; 0-100% per domain of prioritization for (a) life extension, (b) preserving independence, (c) reducing pain and (d) reducing other symptoms)
Co-morbidity | Up to 5 years
  Co-morbidity will be retrieved from the electronic health records (EHR) from the hospital, general practitioner and pharmacy. Data will be registered according to the Charlson' co-morbidity index (CCI; 1-2 mild co-morbidity, 3-4 moderate co-morbidity, 5 severe co-morbidity)
Length-of-stay in hospital/intensive care unit (ICU) | Until hospital discharge, an average of 2 weeks
  Length-of-stay in hospital and on intensive care unit (ICU) in days

SECONDARY OUTCOMES:
Biomarkers | Up to 5 years
  Laboratory values (Hb [mmol/L], leukocytes [/mL), trombocytes [/ml], creatinine [mmol/L], urea [mmol/L], CRP [mg/L], LDL cholesterol [mmol/L], HDL cholesterol [mmol/L], total cholesterol [mmol/L], AST [U/L], ALT [U/L], gGT [U/L], AF [U/L], bilirubin [microl/L], NTproBNP [pg/mL], troponin [microg/L]) will be retrieved from the electronic health records (EHR) from the hospital, general practitioner and pharmacy.
Medication use | Up to 5 years
  Medication use will be retrieved from the electronic health records (EHR) from the hospital, general practitioner and pharmacy.
Treatment (non-pharmacological, including organ support) | Until hospital discharge, up to 3 months
  Treatment (non-pharmacological) will be retrieved from the electronic health records (EHR) from the hospital, general practitioner and (helicopter) emergency medical service. Data will include intravenous fluid resuscitation, vasopressors, mechanical ventilation/non-invasive ventilation, oxygen supply, acute dialysis and extra-corporeal membrane oxygenation (ECMO)
Sequential organ failure assessment (SOFA) | Up to 72 hours after hospitalization
  SOFA scores will be available for patients admitted because of an infection.
Vital parameters | Until hospital discharge, up to 3 months
  Heart rate (bpm), blood pressure (mmHg), oxygen saturation (SpO2, SaO2, PaO2), breathing frequency (per min), consciousness (Glasgow coma scale), pain score (VAS), nausea/vomiting (y/n), defecation (y/n), urination (y/n), body weight (kg), length (cm), fluid balance (ml/day).

CONTACTS AND LOCATIONS:
Overall Officials: Ewoud ter Avest, MD, PhD, Study Chair — University Medical Center Groningen; Jan ter Maaten, MD, PhD, Study Director — University Medical Center Groningen; Hjalmar Bouma, MD, PhD, Study Director — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) may be available to other researchers if needed for their specific research purposes, which amongst others must be in line with the study protocol, the informed consent form and the general data protection regulations (GDPR). Each request for re-use of data will be reviewed by Acutelines' steering group, manager and local review board (LRb), prior to establishing a material and data transfer agreement (MDTA). No IPD will be shared if not required to answer research question.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Supporting information will become available short after initiation of the study and will remain available until the end of the study (undetermined).
Access Criteria: Supporting information will either be made available through the website (http://acutelines.umcg.nl), LinkedIn (https://www.linkedin.com/company/acutelines) and/or upon reasonable request.
URL: http://acutelines.umcg.nl

REFERENCES:
- [Derived] van der Aart TJ, Luxen M, Koeze J, Londen MV, Hackl M, Ter Maaten JC, van Meurs M, Bouma HR; the Acutelines research group. Validation of plasma microRNAs as biomarkers in sepsis associated acute kidney injury upon first clinical presentation reveals limited diagnostic and prognostic performance. PLoS One. 2025 Sep 4;20(9):e0331442. doi: 10.1371/journal.pone.0331442. eCollection 2025. PMID 40906653
- [Derived] van der Aart TJ, Visser M, van Londen M, van de Wetering KMH, Ter Maaten JC, Bouma HR; Acutelines research group. The smell of sepsis: Electronic nose measurements improve early recognition of sepsis in the ED. Am J Emerg Med. 2025 Feb;88:126-133. doi: 10.1016/j.ajem.2024.11.045. Epub 2024 Nov 26. PMID 39615435
- [Derived] Ter Avest E, van Munster BC, van Wijk RJ, Tent S, Ter Horst S, Hu TT, van Heijst LE, van der Veer FS, van Beuningen FE, Ter Maaten JC, Bouma HR. Cohort profile of Acutelines: a large data/biobank of acute and emergency medicine. BMJ Open. 2021 Jul 15;11(7):e047349. doi: 10.1136/bmjopen-2020-047349. PMID 34266842